CLINICAL TRIAL: NCT05321121
Title: Dexmedotomidine for Acute Pain Control in Patients With Multiple Rib Fractures
Brief Title: Dexmedotomidine for Acute Pain Control in Patients With Multiple Rib FracturesRandomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeffrey Nahmias, MD, Associate Professor of Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20216525
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Rib Fractures; Pain, Acute
Keywords: Rib Fracture; Pain; Dexmedotomidine
MeSH Terms: conditions — Rib Fractures; Acute Pain; Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blinded, placebo-controlled trial. Patients will be identified as they present to the trauma bay and meet eligibility criteria. Following informed consent patients will be randomized to either the intervention or control arm. Randomization and allocation concealment will be managed by a nominated independent individual(s) not involved in patient care or data extraction/analysis. The consenting physician will contact the randomization individual by phone. They will use a random number generator to assign group in a 1:1 ratio and then maintain a password protected randomization database that is only accessible to the principal investigator and randomization individual(s).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following informed consent patients will be randomized to either the intervention or control arm. Randomization and allocation concealment will be managed by a nominated independent individual(s) not involved in patient care or data extraction/analysis. The consenting physician will contact the randomization individual by phone. They will use a random number generator to assign group in a 1:1 ratio and then maintain a password protected randomization database that is only accessible to the principal investigator and randomization individual(s).
  The intervention arm will receive an infusion of dexmedetomidine (precedex) at 0.4-0.6 mcg/kg/h (Based off ideal body weight). The control arm will receive an infusion of normal saline. Medication distribution and management will be handled by the Investigational Drug Service (IDS) at UCI medical center. A pharmacist who does not participate in the rest of the study will encode the study drug accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Precedex arm (Experimental): The intervention arm will receive an infusion of dexmedetomidine (precedex) at 0.4-0.6 mcg/kg/h (Based off ideal body weight).
  Interventions: Drug: Dexmedetomidine
- Control arm (Placebo Comparator): The control arm will receive an infusion of normal saline. Medication distribution and management will be handled by the Investigational Drug Service (IDS) at UCI medical center.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedotomidine for Acute Pain Control in Patients with Multiple Rib Fractures
  Arms: Precedex arm
Other: Placebo — The control arm will receive an infusion of normal saline
  Arms: Control arm

SUMMARY:
Blunt chest trauma is the second most common form of unintentional trauma in the US and is associated with significant morbidity and mortality. Thoracic injuries are the third most common cause of death in trauma patients. Rib fractures have an increased associated risk of pneumonia, prolonged hospitalization, and cost. The associated severe pain leads to poor pulmonary mechanics, which contributes to additional complications. Treatment for rib fractures is focused on optimizing analgesia and intense pulmonary hygiene. Most common strategies utilize early mobilization, incentive spirometry (IS), and multimodal pain regimens.

A variety of techniques for analgesia after blunt chest trauma exist. Epidural analgesia is one of the best-studied methods and can often provide significant pain relief. However, this method is invasive, has associated complications, and often can be contraindicated due to coagulopathy or other injuries. Most often a form of multimodal pain strategy is utilized which incorporates acetaminophen, Nonsteroidal anti-inflammatory drugs (NSAIDs), trans-dermal lidocaine, and muscle relaxants. Opioids remain an important adjunct to control severe pain, however, narcotics have their own associated complications.

The aim of our study is to use an infusion of dexmedetomidine (Precedex) to aid in pain management in patients presenting with 3 or more rib fractures. The investigators hypothesize that dexmedetomidine will decrease patient pain and opioid use.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded, placebo-controlled trial. Patients will be identified as they present to the trauma bay and meet eligibility criteria. Following informed consent patients will be randomized to either the intervention or control arm. Randomization and allocation concealment will be managed by a nominated independent individual(s) not involved in patient care or data extraction/analysis. The consenting physician will contact the randomization individual by phone. They will use a random number generator to assign group in a 1:1 ratio and then maintain a password-protected randomization database that is only accessible to the principal investigator and randomization individual(s).

The intervention arm will receive an infusion of dexmedetomidine (precedex) at 0.4-0.6 mcg/kg/h (Based off ideal body weight). The control arm will receive an infusion of normal saline. Medication distribution and management will be handled by the Investigational Drug Service (IDS) at UCI medical center. A pharmacist who does not participate in the rest of the study will encode the study drug accordingly. Dexmedetomidine is approved for ICU and procedural sedation, and its use in this study for analgesics is off-label. A baseline pain assessment will be performed using a numerical pain score (NPS). Infusions will start within 12 hours of arrival to the ICU and will continue for 24 hours. Infusion will stop once the patient is transferred out of the ICU or at 24 hours, whichever is first. In the scenario of possible adverse events (as listed below) the physician can hold or stop the study medication at their discretion. All enrolled patients will also receive a multimodal pain regimen with acetaminophen, NSAIDs, lidocaine patch, gabapentin, and muscle relaxants. For moderate and severe pain (5-10) patients will receive 5-10mg oxycodone every 4-6 hours upon request. Nursing staff will assess pain per the unit standard of care. NPS and opiate administration will be documented in the EMR by the nursing staff. All participants, providers, and staff will be blinded unless medical necessity requires patients to be unblinded.

Data will be collected prospectively from the EMR by blinded researchers and entered into a REDCap database. Data collection will include demographics, mechanism of injury, injury severity score (ISS), imaging, pain scores, pain medications, incentive spirometry, pulmonary complications, ICU LOS, hospital LOS, discharge disposition, and any other clinically relevant data.

Criteria for drop out include:

* Participant withdrawal of consent
* Ordered to drop-out by the investigators or attending physician
* Cases of unmasked blinding

Since both injury severity and age can be confounding variables with pain, the study team plans to do a subgroup analysis after the completion of data collection. Injury severity Score (ISS) ≥ 15 and < 15 will be used to stratify injury severity. Age ≥ 65 and <65 will be used to stratify patient age.

ELIGIBILITY:
Inclusion Criteria:

* Blunt trauma patients
* > 3 rib fractures
* Admission to the ICU

Exclusion Criteria:

Exclusion criteria:

* Younger than 18
* Pregnant
* Prisoners
* History of adverse reaction to dexmedetomidine
* GCS < 14
* Acute CHF exacerbation
* Bradycardia or heart block (HR <55)
* Hypotension (SBP < 90mmHg or MAP < 65mmHg)
* Current opioid use (>30mg OME/day)
* Inability to communicate with staff (dementia)
* Cirrhosis or chronic liver dysfunction (Child Pugh class C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of Pain | through study completion of index hospitalization (up to 6 months)
  Numerical pain score (NPS): a score of 1-10 that will be recorded by the nurse in charge of the patients as standard of care.
Use of morphine and morphine equivalents. | through study completion of index hospitalization (up to 6 months)
  2. Oral morphine equivalents (OME) - A study team member will do a chart review and collect morphine used by the patients.

SECONDARY OUTCOMES:
Epidural administration | through study completion of index hospitalization (up to 6 months)
  Epidural use - patients that fail pain management will be offered an epidural
Time in the hospital | through study completion of index hospitalization (up to 6 months)
  ICU length of stay - number of days in the ICU Hospital length of stay - number of days admitted to the acute care hospital
Respiratory complications | through study completion of index hospitalization (up to 6 months)
  Respiratory complications - include events such as unplanned intubation, pneumonia, pneumothorax and incentive spirometry
Mortality | through study completion of index hospitalization (up to 6 months)
  Mortality - in-hospital mortality rate and 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Nahmias, MD, Principal Investigator — jnahmias@hs.uci.edu
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Lecky FE, Bouamra O, Woodford M, Alexandrescu R, O'Brien SJ. Epidemiology of Polytrauma. In: Damage Control Management in the Polytrauma Patient. New York, NY: Springer New York; 2010:13-24.
- [Background] Carver TW, Kugler NW, Juul J, Peppard WJ, Drescher KM, Somberg LB, Szabo A, Yin Z, Paul JS. Ketamine infusion for pain control in adult patients with multiple rib fractures: Results of a randomized control trial. J Trauma Acute Care Surg. 2019 Feb;86(2):181-188. doi: 10.1097/TA.0000000000002103. PMID 30376537
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Stawicki SP, Grossman MD, Hoey BA, Miller DL, Reed JF 3rd. Rib fractures in the elderly: a marker of injury severity. J Am Geriatr Soc. 2004 May;52(5):805-8. doi: 10.1111/j.1532-5415.2004.52223.x. PMID 15086666
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Result] Gerlach AT, Murphy CV, Dasta JF. An updated focused review of dexmedetomidine in adults. Ann Pharmacother. 2009 Dec;43(12):2064-74. doi: 10.1345/aph.1M310. PMID 19934395
- [Result] Zhang X, Wang D, Shi M, Luo Y. Efficacy and Safety of Dexmedetomidine as an Adjuvant in Epidural Analgesia and Anesthesia: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Clin Drug Investig. 2017 Apr;37(4):343-354. doi: 10.1007/s40261-016-0477-9. PMID 27812971
- [Result] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Result] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Derived] Nahmias J, Stopenski S, Jebbia M, Atallah S, Kirby KA, Alvarez CA, Aryan N, Tay-Lasso E, Dolich M, Lekawa M, Swentek L, Santos J, Schubl S, Kuza C, Nguyen N, Grigorian A. Dexmedetomidine for Analgesia in Nonintubated Patients With Traumatic Rib Fractures: A Randomized Clinical Trial. JAMA Surg. 2025 Oct 1;160(10):1047-1056. doi: 10.1001/jamasurg.2025.3221. PMID 40900569